CLINICAL TRIAL: NCT00030394
Title: A Phase II Study of Gleevec in Ph+ Chronic Phase Chronic Myelogenous Leukemia
Brief Title: Imatinib Mesylate in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01867; AAML0123; U10CA098543 (NIH); CDR0000069161 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Childhood Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who fail to achieve a complete hematologic response after 3 courses or a partial or complete cytogenic response after 6 courses are removed from the study.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying imatinib mesylate to see how well it works in treating patients with chronic myelogenous leukemia. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate in patients with Philadelphia chromosome positive chronic phase chronic myelogenous leukemia treated with imatinib mesylate.

II. Determine the disease-free survival of patients treated with this drug. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine the toxic effects of this drug in these patients. V. Determine the rates of hematological, cytogenetic, and molecular response and time to response in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (chronic myelogenous leukemia [CML] in first chronic phase after failing interferon therapy or demonstrating intolerance to interferon [closed to accrual as of 12/05/03] vs CML relapsing after stem cell transplantation or in second or subsequent chronic phase [closed to accrual as of 7/29/05] vs newly diagnosed CML in first chronic phase with no prior treatment [closed to accrual as of 7/29/05] vs newly diagnosed CML in first chronic phase with no prior treatment).

Patients receive oral imatinib mesylate once daily on days 1-28. Courses repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients who fail to achieve a complete hematologic response after 3 courses or a partial or complete cytogenic response after 6 courses are removed from the study.

PROJECTED ACCRUAL: A total of 109 patients (30 for stratum I [closed to accrual as of 12/05/03] and stratum II [closed to accrual as of 7/29/05], 34 for stratum III [closed to accrual as of 7/29/05], and 45 for stratum IV) will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Philadelphia chromosome positive (Ph+) chronic phase chronic myelogenous leukemia (CML)
* Stratum I (closed to accrual as of 12/05/03):

  * CML in first chronic phase with resistance to interferon alfa (IFN-A) therapy defined as one of the following:

    * WBC count at least 20,000/mm^3 after at least 3 months of treatment with an IFN-A-containing regimen
    * Rising WBC count (at least 100% increase to a level of at least 20,000/mm^3) by two samples at least two weeks apart while receiving treatment with an IFN-A-containing regimen
    * At least 66% Ph+ cells in bone marrow after 1 year of IFN-A therapy
    * At least 30% increase in Ph+ cells in bone marrow after IFN-A-induced cytogenetic response while continuing to receive IFN-A therapy
  * Intolerance to interferon therapy defined as more than two grade 2 toxic effects or any grade 3 toxic effect related to interferon therapy, except grade 3 fever, that is persistent beyond the first 28-day course of therapy and unresponsive to standard supportive care interventions
* Stratum II (closed to accrual as of 7/29/05): CML recurring after stem cell transplantation or in second or subsequent chronic phase

  * No molecular relapse (only evidence is detection of bcr-abl rearrangement with normal bone marrow and blood morphology and normal standard cytogenetic analysis)
* Stratum III (closed to accrual as of 7/29/05): Newly diagnosed CML in first chronic phase with no prior treatment except hydroxyurea
* Stratum IV: Newly diagnosed CML in first chronic phase with no prior treatment except hydroxyurea
* No accelerated or blast phase defined as one or more of the following:

  * WBC doubling time less than 5 days
  * Chloroma
  * Medullary fibrosis
  * More than 10% blasts in peripheral blood or bone marrow
  * More than 20% promyelocytes in peripheral blood or bone marrow
  * More than 20% basophils and eosinophils in peripheral blood
* Performance status - ECOG 0-2
* At least 8 weeks
* See Disease Characteristics
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* Bilirubin no greater than 1.5 times normal
* ALT less than 3.0 times normal
* Albumin greater than 2 g/dL
* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No CNS toxicity greater than grade 2
* See Disease Characteristics
* No prior immunotherapy (for patients in stratum III [closed to accrual as of 7/29/05] and stratum IV only)
* At least 3 months since prior stem cell transplantation (SCT) (patients with allogeneic SCT must have no active graft-versus-host disease [GVHD] and have stable use of steroids) (for patients in stratum II only )
* At least 1 week since prior growth factors
* At least 1 week since prior biologic therapy, including interferon alfa (for patients in stratum I [closed to accrual as of 12/05/03] and stratum II only)
* Recovered from prior immunotherapy
* No concurrent immunomodulating agents
* See Disease Characteristics
* No prior chemotherapy (for patients in stratum III [closed to accrual as of 7/29/05] and stratum IV only)
* At least 6 weeks since prior busulfan or nitrosoureas
* At least 7 days since prior hydroxyurea
* At least 7 days since prior low-dose cytarabine (less than 30 mg/m^2 every 12 to 24 hours)
* At least 14 days since prior moderate-dose cytarabine (100-200 mg/m^2 for 5 to 7 days)
* At least 28 days since prior high-dose cytarabine (1-3 g/m^2 every 12 to 24 hours for 6 to 12 doses)
* At least 21 days since all other cytotoxic chemotherapy
* Recovered from prior chemotherapy
* No concurrent chemotherapy
* No concurrent steroids other than for controlled GVHD in patients with prior allogeneic SCT
* No prior radiotherapy (for patients in stratum III [closed to accrual as of 7/29/05] and stratum IV only)
* At least 2 weeks since prior local palliative (small port) radiotherapy*
* At least 3 months since prior craniospinal radiotherapy or radiotherapy to 50% or more of pelvis*
* At least 6 weeks since prior substantial bone marrow radiotherapy*
* Recovered from prior radiotherapy
* No prior imatinib mesylate
* No concurrent enzyme-activating anticonvulsants
* No concurrent warfarin
* No concurrent naturopathic agents or herbal medicines
* No other concurrent investigational agents
* Concurrent low-molecular weight heparin allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2002-09; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years
Disease-free survival | Up to 5 years
Toxicities graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 5 years

SECONDARY OUTCOMES:
Time to achieve hematological cytogenetic and molecular response | Up to 12 months
  Studied in a multivariate model using a Cox proportional hazards regression model.
Event free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Champagne, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Champagne MA, Fu CH, Chang M, Chen H, Gerbing RB, Alonzo TA, Cooley LD, Heerema NA, Oehler V, Wood C, French ME, Arceci RJ, Smith FO, Bernstein ML. Higher dose imatinib for children with de novo chronic phase chronic myelogenous leukemia: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2011 Jul 15;57(1):56-62. doi: 10.1002/pbc.23031. Epub 2011 Apr 4. PMID 21465636